CLINICAL TRIAL: NCT06076967
Title: Mindfulness Intervention for College Students With ADHD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama, Tuscaloosa (Other)
Collaborators: Wofford College (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GR29540
Record Dates: First submitted 2023-09-25; First posted 2023-10-11 (Actual); Last update posted 2024-08-12 (Actual); Status verified 2024-08

CONDITIONS: Attention Deficit Hyperactivity Disorder
Keywords: ADHD; Mindfulness; College students; Emerging adults
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Acclimatization

STUDY DESIGN:
Intervention Model Description: Students with ADHD will be randomized to a group-based mindfulness intervention or Services-As-Usual (SAU; standard support services provided by the universities).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Adapted Mindful Awareness Practices (MAPS) (Experimental): The Mindful Awareness Practices (MAPs) for ADHD program, an 8-week, group-based mindfulness program for adults with ADHD, has been shown to reduce ADHD, depression, and anxiety symptoms. While promising, it is unknown as to whether the MAPs protocol is feasible, acceptable, and efficacious for college students with ADHD. The current study takes the first step towards enhanced study of mindfulness for college students with ADHD by testing the feasibility, acceptability, and preliminary efficacy of an adapted MAPs protocol delivered within university counseling center settings during the first semester of college.
  Interventions: Behavioral: Mindfulness Awareness Practices for ADHD (adapted)
- Services-As-Usual (Active Comparator): Services-As-Usual includes the standard academic support services provided by university disability/accessibility offices.
  Interventions: Behavioral: Services-As-Usual

INTERVENTIONS:
Behavioral: Mindfulness Awareness Practices for ADHD (adapted) — The Mindful Awareness Practices (MAPs) for ADHD program is an 8-week, group-based mindfulness program for adults with ADHD.
  Arms: Adapted Mindful Awareness Practices (MAPS)
Behavioral: Services-As-Usual — Services-As-Usual includes the standard support services provided by universities
  Arms: Services-As-Usual

SUMMARY:
Attention-deficit/hyperactivity disorder (ADHD) is a neurodevelopmental disorder that commonly persists into adulthood and is associated with significant life impairments. The current study evaluates the feasibility, acceptability, and preliminary efficacy of a group-based mindfulness intervention for first-year college students with ADHD. If found to be feasible, acceptable, and efficacious, subsequent research will examine its impact on a larger scale to have a broader public health impact for college students with ADHD.

DETAILED DESCRIPTION:
Attention-deficit/hyperactivity disorder (ADHD) is a neurodevelopmental disorder that commonly persists into adulthood. Stimulant and non-stimulant pharmacotherapies are the mainstay of treatment; however, non- pharmacological interventions such as mindfulness have significant empirical support. The Mindful Awareness Practices (MAPs) for ADHD program, an 8-week, group-based mindfulness program for adults with ADHD, has been shown to reduce ADHD, depression, and anxiety symptoms. While promising, it is unknown as to whether the MAPs protocol is feasible, acceptable, and efficacious for college students with ADHD. The current study takes the first step towards enhanced study of mindfulness for college students with ADHD by testing the feasibility, acceptability, and preliminary efficacy of an adapted MAPs protocol delivered within university counseling center settings during the first semester of college. First-year college students with ADHD will be recruited at the University of Alabama and Wofford College. After developing and beta testing an adapted MAPs intervention at both sites, students will be randomized to adapted MAPs or Services-As-Usual (SAU; standard support services provided by the universities). Groups will include 10 first-year students and will be run over a 2-year period in the fall semesters (i.e., 4 MAPs groups across the two sites; total MAPs n = 40; total SAU n = 40). MAPs groups will be led by trained therapists in university counseling centers. Assessments will occur at pre, post, and 6-month follow-up using measures of ADHD, sluggish cognitive tempo (SCT), anxiety, and depression symptoms along with emotion regulation and mindfulness, our hypothesized mechanisms of change. Aims of the project are to: 1) adapt, manualize, and beta test the intervention, 2) conduct a pilot randomized controlled trial of adapted MAPs compared to SAU and examine feasibility and acceptability measures and clinical outcomes, and 3) examine whether the adapted MAPs intervention changes the targets hypothesized to be associated with changes in clinical outcomes (i.e., emotional regulation, mindfulness). If adequate feasibility, acceptability, and preliminary efficacy are documented, mindfulness for college students with ADHD can continue to be evaluated in larger trials. If ultimately found to be efficacious, this protocol has the potential to be widely disseminated within college counseling centers to have a broader public health impact for college students with ADHD.

ELIGIBILITY:
Inclusion Criteria:

* First-semester college student with ADHD
* Age 17-25
* Must meet criteria for ADHD
* No major medical problems

Exclusion Criteria:

* Severe depression
* Mania
* Ongoing substance abuse
* Personality disorder that may interfere with group delivery
* Psychotic symptoms
* Recent history of trauma
* Unstable dosage of psychotropic medication

Ages: 17 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-09-15 (Actual); Primary Completion 2026-05-15 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Conners Adult ADHD Rating Scale | Pre-treatment, up to 1-month post-treatment, 6-month follow-up
  This measure assesses adult ADHD symptoms
Adult Concentration Inventory | Pre-treatment, up to 1-month post-treatment, 6-month follow-up
  This measure assesses adult sluggish cognitive tempo (SCT) symptoms
Depression Anxiety Stress Scale-21 | Pre-treatment, up to 1-month post-treatment, 6-month follow-up
  This measure assesses adult anxiety and depression symptoms
Difficulties in Emotion Regulation Scale | Pre-treatment, up to 1-month post-treatment, 6-month follow-up
  This measure assesses emotion regulation abilities in adults.
Trier Social Stress Test | Pre-treatment, up to 1-month post-treatment, 6-month follow-up
  This measure assesses the ability to regulate social stress in a laboratory paradigm.
Mind Excessively Wandering Questionnaire | Pre-treatment, up to 1-month post-treatment, 6-month follow-up
  This measure assesses mind wandering in adults.
Five-Facet Mindfulness Questionnaire | Pre-treatment, up to 1-month post-treatment, 6-month follow-up
  This measure assesses mindfulness in adults.
Sustained Attention to Response Task | Pre-treatment, up to 1-month post-treatment, 6-month follow-up
  This task measures the ability to sustain attention and mind wandering during task performance.
Attention Network Task | Pre-treatment, up to 1-month post-treatment, 6-month follow-up
  This task measures aspects of attention such as alerting, orienting, and executive control.

SECONDARY OUTCOMES:
Behavior Rating Inventory of Executive Function - Adult Version | Pre-treatment, up to 1-month post-treatment, 6-month follow-up
  This measure assesses self-rated executive functioning deficits in adults.
Social Functioning Questionnaire | Pre-treatment, up to 1-month post-treatment, 6-month follow-up
  This measure assesses aspects of social functioning in adults.
Grade Point Average | 6-month follow-up
  This measure assess academic performance in the college setting.

OTHER OUTCOMES:
Treatment Satisfaction and Acceptability Questionnaire | Up to 1-month post-treatment
  This measure will assess participant satisfaction with the treatment.
Session Checklist and Therapist Feedback Form | Weekly during treatment
  This measure will assess whether the therapist delivered each intervention component and will ask the therapist to rate the degree of difficulty with implementation.
Implementation Quality Measure | Weekly sessions will be rated
  This measure will involve a rating of how well the therapist implemented therapy session procedures.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Department of Psychology, University of Alabama, Tuscaloosa, Alabama
  - Department of Psychology, Wofford College, Spartanburg, South Carolina

IPD SHARING:
Plan to Share IPD: Yes
Data will be submitted to the National Institute of Mental Health (NIMH) Data Archive
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will not be released/shared until publication or 12 months after the project end date, whichever comes first.